CLINICAL TRIAL: NCT05888181
Title: Effectiveness and Feasibility of a Mobile Health Self-management Intervention for Patients With Rheumatoid Arthritis: the App-based Education and GOal-setting in Rheumatoid Arthritis Trial
Brief Title: App-based Education and GOal-setting in Rheumatoid Arthritis
Acronym: AEGORA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universitaire Ziekenhuizen KU Leuven (Other)
Collaborators: Sidekick Health (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: S66633
Record Dates: First submitted 2023-03-23; First posted 2023-06-05 (Actual); Results first posted 2025-05-16 (Actual); Last update posted 2025-05-16 (Actual); Status verified 2023-05

CONDITIONS: Rheumatoid Arthritis
Keywords: self-management; mobile health; smartphone applications; education; patient-reported outcomes; lifestyle; goal-setting; remote monitoring
MeSH Terms: conditions — Arthritis, Rheumatoid

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Intervention group A (weekly RAID) (Experimental): Access to the study app with weekly prompts to complete the patient-reported questionnaire Rheumatoid Arthritis Impact of Disease (RAID)
  Interventions: Other: Mobile app-based self-management intervention
- Intervention group B (monthly RAID) (Experimental): Access to the study app with monthly prompts to complete the patient-reported questionnaire Rheumatoid Arthritis Impact of Disease (RAID)
  Interventions: Other: Mobile app-based self-management intervention
- Control group (usual care) (No Intervention): No access to the study app, follow-up according to usual care standards. This includes informal screening for general wellbeing during outpatient clinic visits, with referral to specific allied health professionals for additional education or non-pharmacological support if needed. The scores derived from study-related questionnaires can be used as a guide for these discussions. As part of standard care, participants in both the control group and the intervention groups will also receive a standardised educational leaflet about RA.

INTERVENTIONS:
Other: Mobile app-based self-management intervention — The self-management program, accessible via a smartphone app, comprises several components. First, the app contains an RA-specific educational program presented as videos in 16 weekly modules. Second, the app provides patients with tailored lifestyle advice, both as part of the educational program and in the form of personalized messages from a certified health coach. Third, the study app includes remote monitoring features underpinned by goal-setting principles. For instance, participants can use the app to log daily steps and physical activity, as well as their diet, sleep, and mental health. Personal goals, as well as physical challenges and meditation or mindfulness exercises, can be set up within the app to encourage behavioral change.
  Finally, patient-reported disease burden can be monitored within the study app via the RAID instrument. Based on random allocation to one of both intervention groups, the RAID will be prompted either weekly (group A) or monthly (group B).
  Arms: Intervention group A (weekly RAID); Intervention group B (monthly RAID)

SUMMARY:
The purpose of this pragmatic, investigator-initiated, multicentre randomised controlled trial is to study the effectiveness and feasibility of a mobile app-based self-management intervention for patients with rheumatoid arthritis (RA), aiming to improve self-efficacy for the management of RA-related symptoms. The intervention consists of education, lifestyle advice and remote monitoring elements and is based on principles of goal setting, self-efficacy theory and behavioural economics, embedded within a platform supported by motivational features and gamification. The primary endpoint is defined as achieving at least a minimal clinically important difference in arthritis-related self-efficacy (the ASES-score) at the follow-up visit in favour of the intervention group when compared to the control group.

Moreover, although qualitative studies have highlighted concerns among both patients and healthcare professionals that mobile apps might induce illness behaviour by increasing patients' awareness of their symptoms, this has rarely been studied in detail. Consequently, data regarding the effects of remote monitoring on symptom hypervigilance remain limited and conflicting. Therefore, this trial additionally aims to assess (as a key secondary objective) if a mobile app-based intervention is associated with changes in pain catastrophising, as a conceptualisation of hypervigilance to symptoms.

ELIGIBILITY:
Patients will be considered eligible for participation in the study if they:

* Are able and willing to provide written informed consent for participation.
* Are 18 years of age or older.
* Have a diagnosis of RA made by a rheumatologist, with a minimal time since diagnosis of 16 weeks. This time frame was chosen based on conceptual reasons and previous work of our research group, suggesting that the dynamic and impactful first weeks after diagnosis are not the ideal time window to assess psychosocial outcomes.
* Are able to understand and read Dutch.
* Have access to a smartphone that meets the technical requirements to run the study application, including an Android (8.0 or more recent) or Apple iOS (14.0 or more recent) operating system, and feel comfortable using it.

In order to include an optimally representative patient population, no additional exclusion criteria will be applied for this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 128 (Actual)
Dates: Start 2023-03-03 (Actual); Primary Completion 2024-02-06 (Actual); Study Completion 2024-02-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Patrick Verschueren, MD, PhD, Principal Investigator — University Hospitals KU Leuven
Locations (2):
- Belgium (2):
  - UZ Leuven, Leuven, Vlaams Brabant
  - AZ Sint-Lucas Brugge, Bruges, West-Vlaanderen

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Doumen M, Westhovens R, Pazmino S, Bertrand D, Stouten V, Neys C, Creten N, Van Laeken E, Verschueren P, De Cock D. The ideal mHealth-application for rheumatoid arthritis: qualitative findings from stakeholder focus groups. BMC Musculoskelet Disord. 2021 Aug 30;22(1):746. doi: 10.1186/s12891-021-04624-8. PMID 34461875
- [Background] Doumen M, De Cock D, Van Lierde C, Betrains A, Pazmino S, Bertrand D, Westhovens R, Verschueren P. Engagement and attrition with eHealth tools for remote monitoring in chronic arthritis: a systematic review and meta-analysis. RMD Open. 2022 Oct;8(2):e002625. doi: 10.1136/rmdopen-2022-002625. PMID 36302561
- [Background] Van der Elst K, Mathijssen EGE, Landgren E, Bremander A, De Groef A, Lindqvist E, Nylander M, Peters A, Van den Hoogen F, van Eijk-Hustings Y, Verhoeven G, Vriezekolk JE, Westhovens R, Larsson I. What do patients prefer? A multinational, longitudinal, qualitative study on patient-preferred treatment outcomes in early rheumatoid arthritis. RMD Open. 2020 Sep;6(2):e001339. doi: 10.1136/rmdopen-2020-001339. PMID 32938747
- [Background] Van der Elst K, Verschueren P, De Cock D, De Groef A, Stouten V, Pazmino S, Vriezekolk J, Joly J, Moons P, Westhovens R. One in five patients with rapidly and persistently controlled early rheumatoid arthritis report poor well-being after 1 year of treatment. RMD Open. 2020 Apr;6(1):e001146. doi: 10.1136/rmdopen-2019-001146. PMID 32371432
- [Background] Doumen M, De Cock D, Pazmino S, Bertrand D, Joly J, Westhovens R, Verschueren P. Psychosocial Burden Predicts Sustained Remission in Early Rheumatoid Arthritis: Unraveling the Complex Interplay of Well-Being and Disease Activity. Arthritis Care Res (Hoboken). 2023 Apr;75(4):758-767. doi: 10.1002/acr.24847. Epub 2022 Nov 28. PMID 34931480
- [Background] Doumen M, De Cock D, Pazmino S, Bertrand D, Joly J, Westhovens R, Verschueren P. Treatment response and several patient-reported outcomes are early determinants of future self-efficacy in rheumatoid arthritis. Arthritis Res Ther. 2021 Oct 27;23(1):269. doi: 10.1186/s13075-021-02651-3. PMID 34706771
- [Background] Doumen M, Pazmino S, Bertrand D, De Cock D, Joly J, Westhovens R, Verschueren P. Longitudinal trajectories of fatigue in early RA: the role of inflammation, perceived disease impact and early treatment response. Ann Rheum Dis. 2022 Oct;81(10):1385-1391. doi: 10.1136/annrheumdis-2022-222517. Epub 2022 Jun 20. PMID 35725296
- [Background] Doumen M, De Meyst E, Lefevre C, Pazmino S, Joly J, Bertrand D, Devinck M, Westhovens R, Verschueren P. Effectiveness and feasibility of a mobile health self-management intervention in rheumatoid arthritis: study protocol for a pragmatic multicentre randomised controlled trial (AEGORA). Trials. 2023 Oct 28;24(1):697. doi: 10.1186/s13063-023-07733-y. PMID 37898781
- [Derived] Doumen M, De Meyst E, Bertrand D, Pazmino S, Piessens M, Joly J, Devinck M, Westhovens R, Verschueren P. A mobile app to support self-management and remotely monitor disease impact in rheumatoid arthritis: the randomized controlled AEGORA trial. Rheumatology (Oxford). 2025 May 1;64(5):2505-2514. doi: 10.1093/rheumatology/keae638. PMID 39576683

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Of 128 enrolled participants, 122 completed the necessary baseline assessments and installed the study app. These were entered in the ITT population.
Groups:
- Intervention Group A (Weekly RAID): Access to the study app with weekly prompts to complete the patient-reported questionnaire Rheumatoid Arthritis Impact of Disease (RAID)
  Mobile app-based self-management intervention: The self-management program, accessible via a smartphone app, comprises several components. First, the app contains an RA-specific educational program presented as videos in 16 weekly modules. Second, the app provides patients with tailored lifestyle advice, both as part of the educational program and in the form of personalized messages from a certified health coach. Third, the study app includes remote monitoring features underpinned by goal-setting principles. For instance, participants can use the app to log daily steps and physical activity, as well as their diet, sleep, and mental health. Personal goals, as well as physical challenges and meditation or mindfulness exercises, can be set up within the app to encourage behavioral change.
  Finally, patient-reported disease burden can be monitored within the study app via the RAID instrument. Based on random allocation to one of both intervention groups, the RAID will be prompted either weekly (group A) or monthly (group B).
- Intervention Group B (Monthly RAID): Access to the study app with monthly prompts to complete the patient-reported questionnaire Rheumatoid Arthritis Impact of Disease (RAID)
  Mobile app-based self-management intervention: The self-management program, accessible via a smartphone app, comprises several components. First, the app contains an RA-specific educational program presented as videos in 16 weekly modules. Second, the app provides patients with tailored lifestyle advice, both as part of the educational program and in the form of personalized messages from a certified health coach. Third, the study app includes remote monitoring features underpinned by goal-setting principles. For instance, participants can use the app to log daily steps and physical activity, as well as their diet, sleep, and mental health. Personal goals, as well as physical challenges and meditation or mindfulness exercises, can be set up within the app to encourage behavioral change.
  Finally, patient-reported disease burden can be monitored within the study app via the RAID instrument. Based on random allocation to one of both intervention groups, the RAID will be prompted either weekly (group A) or monthly (group B).
Period: Overall Study
Arm/Group | Intervention Group A (Weekly RAID) | Intervention Group B (Monthly RAID) | Control Group (Usual Care)
Started | 30 | 30 | 62
Completed | 29 | 29 | 62
Not Completed | 1 | 1 | 0
Not completed — Lost to Follow-up | 1 | 1 | 0

BASELINE CHARACTERISTICS:
Population: For baseline characteristics and primary analyses, intervention groups A and B were combined (as predefined in the protocol).
Groups:
- Combined Intervention Group (A & B): Access to the study app with either weekly or monthly prompts to complete the patient-reported questionnaire Rheumatoid Arthritis Impact of Disease (RAID)
  Mobile app-based self-management intervention: The self-management program, accessible via a smartphone app, comprises several components. First, the app contains an RA-specific educational program presented as videos in 16 weekly modules. Second, the app provides patients with tailored lifestyle advice, both as part of the educational program and in the form of personalized messages from a certified health coach. Third, the study app includes remote monitoring features underpinned by goal-setting principles. For instance, participants can use the app to log daily steps and physical activity, as well as their diet, sleep, and mental health. Personal goals, as well as physical challenges and meditation or mindfulness exercises, can be set up within the app to encourage behavioral change.
  Finally, patient-reported disease burden can be monitored within the study app via the RAID instrument. Based on random allocation to one of both intervention groups, the RAID will be prompted either weekly (group A) or monthly (group B).
- Total: Total of all reporting groups
Arm/Group | Combined Intervention Group (A & B) | Control Group (Usual Care) | Total
Number analyzed (Participants) | 60 | 62 | 122
Age, Continuous [Mean (Standard Deviation); unit: years] | 58 (12) | 58 (11) | 58 (12)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 38 | 45 | 83
  Male | 22 | 17 | 39
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
RF/ACPA positive [Count of Participants; unit: Participants] | 43 | 55 | 98
Erosive disease [Count of Participants; unit: Participants] | 26 | 27 | 53
Disease duration, years [Mean (Standard Deviation); unit: years] | 11 (9) | 13 (10) | 12 (10)
BMI [Mean (Standard Deviation); unit: kg/m2] | 26 (5) | 27 (5) | 27 (5)
Smoking ever [Count of Participants; unit: Participants] | 30 | 27 | 57
Rheumatic Disease Comorbidity Index (RDCI) [Mean (Standard Deviation); unit: units on a scale] | 1.1 (1.4) | 1.5 (1.5) | 1.3 (1.5)
DAS28-CRP [Mean (Standard Deviation); unit: units on a scale] | 2.3 (0.9) | 2.4 (1.0) | 2.4 (1.0)
Health Assessment Questionnaire (HAQ) [Mean (Standard Deviation); unit: units on a scale] | 0.7 (0.7) | 0.6 (0.6) | 0.6 (0.6)
Rheumatoid Arthritis Impact of Disease (RAID) [Mean (Standard Deviation); unit: units on a scale] | 3.6 (2.4) | 3.7 (2.3) | 3.7 (2.4)
Arthritis Self-Efficacy Scale (ASES) [Mean (Standard Deviation); unit: units on a scale] | 72 (22) | 72 (20) | 72 (22)
Pain Catastrophizing Scale (PCS) [Mean (Standard Deviation); unit: units on a scale] | 13 (11) | 14 (13) | 14 (13)

OUTCOME MEASURES:

1. Primary Outcome: Arthritis Self-Efficacy Scale (ASES)
Description: Superiority outcome. The ASES is a patient-reported questionnaire consisting of 20 items across 2 subscales: self-efficacy for managing pain (range 5-50), and self-efficacy for controlling other symptoms (range 6-60). Both scores can be summed to derive a total ASES-score (range 11-110). Higher scores indicate higher perceived self-efficacy.
Time Frame: At follow-up visit (4-6 months from baseline)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Combined Intervention Group (A & B) | Control Group (Usual Care)
Number analyzed (Participants) | 60 | 62
score on a scale | 74 (22) | 74 (20)

2. Secondary Outcome: Pain Catastrophizing Scale (PCS)
Description: Non-inferiority outcome. The PCS comprises 13 items on a 0-4 Likert scale, resulting in a total score of 0-52 with subscales for rumination, magnification, and helplessness. Higher scores indicate more catastrophic perceptions concerning pain.
  Additionally, a post-hoc analysis will be carried out comparing the PCS between intervention group A and B, to study the influence of PRO-reporting frequency on pain catastrophising.
Time Frame: At follow-up visit (4-6 months from baseline)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Combined Intervention Group (A & B) | Control Group (Usual Care)
Number analyzed (Participants) | 60 | 62
score on a scale | 11 (8) | 13 (10)

3. Secondary Outcome: Rheumatoid Arthritis Impact of Disease (RAID)
Description: Superiority outcome. The RAID consists of 7 items on a 0-10 numeric rating scale, enquiring about the impact of RA on pain, functional limitations, fatigue, sleep, physical wellbeing, emotional wellbeing, and coping. A total RAID score (0-10) is derived as a weighted average of the 7 subscores (Pain: 21%, Functional disability: 16%, Fatigue: 15%, Emotional well-being: 12%, Sleep: 12%, Coping: 12%, Physical well-being: 12%). Higher scores on both the total scale and the subscales indicate more perceived disease impact.
Time Frame: At follow-up visit (4-6 months from baseline)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Combined Intervention Group (A & B) | Control Group (Usual Care)
Number analyzed (Participants) | 60 | 62
score on a scale | 3.6 (2.4) | 3.5 (2.2)

4. Secondary Outcome: International Physical Activity Questionnaire Short Form (IPAQ-S)
Description: Superiority outcome. The IPAQ-S is a 7-item questionnaire enquiring about physical activities during the last 7 days. An activity score is obtained for different domains, each multiplied with the accompanying metabolic equivalent of task (MET) value, leading to a sum score corresponding with low, moderate, or high physical activity.
Time Frame: At follow-up visit (4-6 months from baseline)
Measure: Mean (Standard Deviation); unit: MET minutes/week
Arm/Group | Combined Intervention Group (A & B) | Control Group (Usual Care)
Number analyzed (Participants) | 60 | 62
MET minutes/week | 5036 (3927) | 4674 (4046)

5. Secondary Outcome: Pittsburgh Sleep Quality Index (PSQI)
Description: Superiority outcome. The PSQI measures sleep quality through 19 items across 7 domains, with a resulting total score ranging from 0-21.Higher scores indicate worse sleep quality.
Time Frame: At follow-up visit (4-6 months from baseline)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Combined Intervention Group (A & B) | Control Group (Usual Care)
Number analyzed (Participants) | 60 | 62
score on a scale | 7.5 (3.9) | 8.0 (3.6)

6. Other Pre Specified Outcome: Participant Engagement With Study Application: Remote Monitoring of RAID
Description: The proportion of in-app completed RAID questionnaires will be calculated as the ratio (%) between completed questionnaires and the total number of questionnaires that were prompted throughout the study period.
Time Frame: Throughout study period (intervention arms only): 4-6 months. Specifically, these data will be collected at the follow-up visit (4-6 months from baseline) and reported for the whole study period.
Measure: Number; unit: percentage completed RAIDs
Arm/Group | Intervention Group A (Weekly RAID) | Intervention Group B (Monthly RAID)
Number analyzed (Participants) | 30 | 30
percentage completed RAIDs | 47 | 53

7. Other Pre Specified Outcome: Participant Engagement With Study Application: Usage of the App
Description: Usage data will be logged passively in the study app. Usage data consist of information concerning how often the app and its core functions are accessed. Specifically, we will calculate the proportion of days where the study app was accessed, and the proportion of days where an educational video was viewed within the study app.
Time Frame: as for outcome 6
Reporting Status: Not Posted

8. Other Pre Specified Outcome: Participant Engagement With Study Application: Daily Step Count
Description: When users choose to activate this function, the number of steps per day will also be passively logged in the study app. When available, we will analyze daily step patterns descriptively (proportion meeting the WHO-recommended daily target, evolution over time, correlation with IPAQ-S score, and correlation with symptoms based on the RAID).
Time Frame: as for outcome 6
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: 4-6 months (duration of the study)
Arm/Group | Intervention Group A (Weekly RAID) | Intervention Group B (Monthly RAID) | Control Group (Usual Care)
All-Cause Mortality (participants affected / at risk) | 0/30 | 0/30 | 0/62
Serious Adverse Events (participants affected / at risk) | 0/30 | 0/30 | 0/62
Other Adverse Events (participants affected / at risk) | 0/30 | 0/30 | 0/62

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-11-03): https://cdn.clinicaltrials.gov/large-docs/81/NCT05888181/Prot_SAP_000.pdf